CLINICAL TRIAL: NCT06040931
Title: Relationship Between Airway Inflammation, Small Airways Dysfunction, and Frequency of Acute Exacerbations in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Airway Inflammation, Small Airways Dysfunction, and Frequency of Exacerbations in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Collaborators: Azza Tarik Eliwa (Unknown); Ahmed Elsayed Mansour (Unknown); Taha Taha Abdelgawad (Unknown); Ahmed Mohamed Fouda (Unknown)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Assistant lecturer, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: M.S.21.08.1628
Record Dates: First submitted 2023-09-07; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: COPD Exacerbation Acute
Keywords: neutrophilic airway inflammation; small airways dysfunction; acute exacerbation; stable COPD patients
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Intervention Model Description: prospective correlational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrequent exacerbators (IFE) group (Active Comparator): 15 patients with infrequent exacerbation (IFE) "≤1 exacerbation per year in the preceding 12 months before enrolment.
  Interventions: Procedure: Bronchoscopy
- Frequent exacerbators (FE) group (Active Comparator): 15 patients with frequent exacerbation(FE) "≥ 2 per year in the preceding 12 months before enrolment
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy and broncho-alveolar lavage (BAL) to assess neutrophilic count in BAL as a measurement of airway inflammation
  Other Names: body Plethysmography (RV/TLC); Spirometry "pre and post bronchdilator to show poorly reversible airway obstruobstructin; CT-chest (Paired Inspiratory and expiratory HRCT scan) and measuring mean lung density

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common, preventable, and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases Chronic Obstructive Pulmonary Disease (COPD) is a heterogenous disease of the lungs that can comprise of different pathophysiological phenotypes, including emphysema, chronic bronchitis, and Small Airways Disease (SAD). COPD is also associated with chronic inflammation and this ongoing inflammation may result in airway remodeling and excessive mucus plugging within the small airways Small airways disease (SAD) is a cardinal feature of chronic obstructive pulmonary disease (COPD) first recognized in the nineteenth century. The diverse histopathological features associated with SAD underpin the heterogeneous nature of COPD. The small airways have been defined as < 2mm diameter and arise from the 4th - 13th generation of airway branching (taking trachea as 1st generation to alveoli as 23rd), but on average arise by the 8th aim of this work is to study the relationship between neutrophilic airway inflammation, small airways dysfunction, and frequency of acute exacerbation in stable COPD patients

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common, preventable, and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases Chronic Obstructive Pulmonary Disease (COPD) is a heterogenous disease of the lungs that can comprise of different pathophysiological phenotypes, including emphysema, chronic bronchitis, and Small Airways Disease (SAD). COPD is also associated with chronic inflammation and this ongoing inflammation may result in airway remodeling and excessive mucus plugging within the small airways Small airways disease (SAD) is a cardinal feature of chronic obstructive pulmonary disease (COPD) first recognized in the nineteenth century. The diverse histopathological features associated with SAD underpin the heterogeneous nature of COPD. The small airways have been defined as < 2mm diameter and arise from the 4th - 13th generation of airway branching (taking trachea as 1st generation to alveoli as 23rd), but on average arise by the 8th Small airway disease (SAD) has been recognized for many years as a central feature of chronic obstructive pulmonary disease (COPD). Histopathology studies have shown that the narrowing and destruction of small airways in COPD combined with inflammatory cell infiltration in the submucosa increases the severity of the disease. SAD is present in the early stages of COPD and becomes more widespread over time as the disease progresses to more severe COPD Exacerbations are an acute worsening of symptoms resulting in additional therapy and can be classified as mild, moderate, or severe, Exacerbations are associated with faster lung function decline and hospital admissions During both stable periods and exacerbations, there is increased neutrophilic inflammation in the airways of COPD subjects , Neutrophilic inflammation is a common feature of many airway diseases and is associated with disease progression, often irrespective of the initiating cause or underlying diagnosis The aim of this work is to study the relationship between neutrophilic airway inflammation, small airways dysfunction, and frequency of acute exacerbation in stable COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of COPD according to GOLD 2021
* Patients should quit smoking at least 6 months before enrolment in the study.

Exclusion Criteria:

* Pulmonary diseases other than COPD e.g parenchymatous lung diseases
* Active smokers.
* Patients unfit for bronchoscopy.
* Immunosuppressive state and immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation between neutrophilic airway inflammation and stable COPD patients | one year
  Concentration of neutrophilic count (cell/ml)in BAL
Correlation between frequency of acute exacerbation and stable COPD patients | One year
  Rate of exacerbation / year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, lecturer, Principal Investigator — Mansoura university Faculty of medicine
Locations (1):
- faculty of medicine Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No